CLINICAL TRIAL: NCT07057297
Title: Residual Stenosis and Restenosis Following Carotid Endarterectomy With Primary Closure, A Prospective Tracking Study
Acronym: RECEPT
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Collaborators: The University Hospital Plzeň (Unknown); Masaryk Hospital Usti nad Labem (Other); University Hospital Olomouc (Other); County Hospital Liberec, Liberec, Czech Republic (Unknown)
Responsible Party: Principal Investigator, Norbert Svoboda, cpt. MD. Norbert Svoboda, PhD., FEBNS, Charles University, Czech Republic
Other Study IDs: 108/19-31/2024
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Carotid Arteriosclerosis; Carotid Stenosis; Brain Stroke
Keywords: Carotid Artery; Atherosclerosis; Endarterectomy; Stroke
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Atherosclerosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients after carotid endarterectomy: Included paitnets with sign informed consent after carotid endarterectomy

SUMMARY:
This prospective, multicenter observational study aims to evaluate the incidence, timing, and characteristics of residual and recurrent (restenosis) carotid artery stenosis following carotid endarterectomy (CEA) with primary closure. Conducted across several neurosurgical centers in the Czech Republic, the study will include patients undergoing elective CEA who meet standard clinical indications.

Participants will undergo preoperative CT angiography and follow-up imaging at 30 days and 1 year post-surgery. Residual stenosis is defined as ≥50% luminal narrowing detected within 30 days postoperatively, while restenosis is evaluated at later time points. The study will also assess clinical outcomes such as ischemic stroke, TIA, myocardial infarction, and mortality. The standardized surgical technique and harmonized diagnostic algorithm across all centers aim to provide robust data on the performance and durability of primary closure CEA.

DETAILED DESCRIPTION:
Study Objective:

The objective of this study is to assess the true incidence of restenosis following CEA in the Czech Republic. A major advantage of this study is the use of standardized surgical procedures across participating centers, along with unified data collection methods and diagnostic algorithms.

Methodology:

Patient Cohort:

All patients meeting the current guideline indications for CEA will be enrolled.

Exclusion criteria include:

Age ≤18 or ≥90 years

Previous endarterectomy or stenting

Unsuitable vascular anatomy

High perioperative risk

Contralateral cranial nerve X or XII palsy

History of neck irradiation

Tandem carotid stenosis or intracranial vascular pathology (e.g., aneurysm or AVM)

Absence of signed informed consent

Collected data will include:

Epidemiologic risk factors: age, sex, diabetes, hypertension, dyslipidemia, metabolic syndrome, renal insufficiency, smoking, physical activity, weight, comorbidities

Laboratory markers: LDL, HDL, cholesterol, lipoprotein A, triglycerides, CKD-EPI, sedimentation rate, fibrinogen, INR (Quick test), APTT

Diagnostics:

All patients will undergo non-contrast brain CT. Carotid stenosis will be assessed by CT angiography performed within 3 months prior to surgery. In addition to stenosis severity, the degree of calcification will be classified as:

No calcification

Minimal

Partially calcified

Pronounced

Severe/unable to evaluate

Other vascular pathology will also be recorded. Follow-up imaging will be performed at 1 month and 1 year postoperatively. CT findings will be assessed by two independent reviewers.

Surgical Technique:

All patients will receive mono- or dual antiplatelet therapy, and 5,000 IU of heparin will be administered intraoperatively. Surgery may be performed under general anesthesia with electrophysiological monitoring or under local anesthesia, based on the surgeon's preference.

A longitudinal incision will be made anterior to the sternocleidomastoid muscle. The common carotid artery and its branches will be dissected and clamped. The internal carotid artery will be clamped distal to the most significant stenosis, as identified on preoperative CTA. The surgeon will incise through the tunica adventitia and media to expose and excise the atherosclerotic plaque. Any residual fragments will be removed, and the arterial wall will be closed using 6/0 suture.

Follow-Up:

Patients will continue on mono- or dual antiplatelet therapy. Mandatory follow-up CT angiography will be performed at 30 days and1 year. During follow-up, the following will be evaluated:

CTA findings

Overall patient condition

Incidence of ischemic stroke (iCMP), TIA, myocardial infarction, and death

Outcomes:

Primary Outcome:

Restenosis ≥50% at 12 months

Secondary Outcomes:

Residual stenosis ≥50% at 30 days

iCMP/TIA/death/MI

Change in modified Rankin Scale (mRS)

Timeline:

All participating centers (ÚVN, ČB, ÚNL, Poruba, Plzeň, Liberec, Zlín, Olomouc, Hradec Králové, Fifejdy, Ostrava) together treat approximately 600-700 patients annually.

An estimated 350 patients will be enrolled within 6 months. By the end of 2026, 300 patients will be included (expected dropout: 50).

This will allow evaluation of:

Secondary outcomes in all 300 patients

Primary outcome in approximately 8 out of 26 centers (those with complete 12-month data)

Ethical Approval:

All participating centers have received approval from their respective institutional ethics committees.

Funding:

This study is conducted without external financial support.

ELIGIBILITY:
Inclusion Criteria:

Patients without matching any of exclusion criteria who underwent cartotid endarterectomy

Exclusion Criteria:

Age ≤18 or ≥90 years

Previous endarterectomy or stenting

Unsuitable vascular anatomy

High perioperative risk

Contralateral cranial nerve X or XII palsy

History of neck irradiation

Tandem carotid stenosis or intracranial vascular pathology (e.g., aneurysm or AVM)

Absence of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo carotid endarterectomy for carotid artery stenosis with primary suture.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Restenosis ≥50% at 12 months | 12 months
  Restenosis ≥50% at 12 months

SECONDARY OUTCOMES:
Restenosis ≥50% | 30 days
  Restenosis ≥50%
iCMP/TIA/death/MI | 1 year
  iCMP/TIA/death/MI
Change in modified Rankin Scale (mRS) | 1 year
  Change in modified Rankin Scale (mRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Central Military Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Epidemiologic risk factors: age, sex, diabetes, hypertension, dyslipidemia, metabolic syndrome, renal insufficiency, smoking, physical activity, weight, comorbidities
  Laboratory markers: LDL, HDL, cholesterol, lipoprotein A, triglycerides, CKD-EPI, sedimentation rate, fibrinogen, INR (Quick test), APTT
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2/2027 - 2/2028
Access Criteria: online

DOCUMENTS (1):
  • Study Protocol (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/97/NCT07057297/Prot_000.pdf